CLINICAL TRIAL: NCT04438356
Title: Effects of Mobile Health Care for Patients After Acute Myocardial Infarction on Disease Perception, Self-Efficacy, Anxiety and Cardio-Respiratory Fitness: A Randomized Controlled Trial
Brief Title: M-Health Care for Patients After AMI on Disease Perception, Self-Efficacy, Anxiety and Cardio-Respiratory Fitness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Hui-Hsun Chiang, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: M-Health Care for AMI Patients
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Mobile Health; Acute Myocardial Infarction; Undefined; Self-efficacy; Anxiety; Cardio-respiratory Fitness
Keywords: Mobile Health; self-efficacy; disease perception; Anxiety; cardio-respiratory fitness; Remote Care
MeSH Terms: conditions — Anxiety Disorders | interventions — American Recovery and Reinvestment Act

STUDY DESIGN:
Intervention Model Description: wait list control group RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-health (Experimental): After the acute myocardial infarction, patients will be randomly assigned to the intervention group. Give the intervention group mobile health care programs and given Garmin monitoring hands ring. In order to give patients clear walking goals and exercise intensity, the intervention group will use the Mobile Health Medical Line app to remind patients of the walking frequency and time, and use Garmin monitoring bracelet to record the patient's daily walking steps. The Mobile Health Medical Line app content includes: 1. Encourage the walking exercise to perform 2. Give them knowledge about acute myocardial infarction 3. How to self-care themselves 4. How to release their anxiety?
  Interventions: Combination Product: M-Health
- wait list control (Experimental): wait list control for 3 months and then use the Mobile Health Medical Line app to remind patients of the walking frequency and time, and use Garmin monitoring bracelet to record the patient's daily walking steps. The Mobile Health Medical Line app content includes: 1. Encourage the walking exercise to perform 2. Give them knowledge about acute myocardial infarction 3. How to self-care themselves 4. How to release their anxiety?
  Interventions: Combination Product: M-Health

INTERVENTIONS:
Combination Product: M-Health — The study was randomized (wait-list-control), and it was estimated that 80 subjects were randomly assigned to the immediate treatment group and the wait-list-control group. The two groups were tested for baseline before intervention in the mHealth. After the first questionnaire evaluation, the experimental group was involved in the mHealth for three months, and after three months, the experimental group and the waiting intervention control group were post-tested. To assess the effectiveness of the two groups before and after the mHealth . Control group that waits for intervention in the fourth month from the beginning of the fourth month to the end of the sixth month.

SUMMARY:
The aim of this study is to explore the overall effectiveness of interventions using mobile health care to improve disease perception, self-efficacy, anxiety, cardio-pulmonary fitness for patients with acute myocardial infarction.

DETAILED DESCRIPTION:
Heart disease is the second leading cause of death in Taiwan. Coronary artery disease (CAD) is the majority, and coronary artery disease is the most common cardiovascular disease. There is an increase, and it is no longer just that the elderly is the predominant group. There is a tendency to gradually become younger. In foreign countries, coronary heart disease is also one of the main causes of patient death and disability, resulting in huge medical burdens and costs. Coronary heart disease also includes acute myocardial infarction, which causes myocardial cell death due to unstable myocardial ischemia. Sudden heart disease brings unexpected shock, fear, and despair to patients and their families. Therefore, patient self-management is very important. It also improves the patient's quality of life.

Post-acute myocardial infarction patients are susceptible to piecemeal information and lack the motivation to change their life style, continue to maintain smoking behavior and do not engage in exercise, leading to the recurrence of major coronary artery problems. In order to reduce secondary cardiovascular problems, it is necessary to rely on the patient's own knowledge of the disease, self-care behavior and self-efficacy, including diet, exercise, etc., so that the disease can be controlled and treated, and also need to monitor and adjust the physical and mental state to reduce subsequent problems caused by anxiety. Therefore, in order to provide multi-party support for patients' self-health care, mobile health care such as mobile phone text messages, applications, and remote monitoring are gradually emerging. Therefore, it is expected that the use of mHealth can be used to develop two-way communication and interaction and a higher message reception rate to stimulate acuteness. After myocardial infarction, patients can change their motivations for self-health care behaviors to achieve more efficient disease perception, self-efficacy, anxiety and cardiopulmonary fitness, and have a longer-term influence ability.

ELIGIBILITY:
Inclusion Criteria:

* Taiwanese, understand Chinese
* Patients who are over 20 years old and have AMI (including ST segment ascending and non-ST segment ascending), diagnosed by percutaneous coronary intervention and without complications within 30±5 days, the left ventricular injection rate is greater than 40% .
* Ability and willingness to provide informed consent.
* Have a smartphone.
* Can receive and send smartphone messages.

Exclusion Criteria:

* Those who can't express their wishes clearly (such as mental dysfunction)
* mental disorder
* Patients who participate in other research projects
* Planned coronary artery bypass surgery or other diseases that require continuous heart care.
* Abuse of alcohol or narcotics.
* Left ventricular ejection fraction (LVEF) is less than 40%.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Disease Perception-T1 | T1-baseline
  The Brief Illness Perception Questionnaire(The B-IPQ) have nine questions on the scale. The first eight questions use a response level of 0 to 10. The ninth question is an open question and answer. The patient is asked to list the three most important causes of the disease. The higher the total score, the greater the threat to the disease.
Disease Perception-T2 | T2-three months later
  The Brief Illness Perception Questionnaire(The B-IPQ) have nine questions on the scale. The first eight questions use a response level of 0 to 10. The ninth question is an open question and answer. The patient is asked to list the three most important causes of the disease. The higher the total score, the greater the threat to the disease.
Disease Perception-T3 | T3-six months later
  The Brief Illness Perception Questionnaire(The B-IPQ) have nine questions on the scale. The first eight questions use a response level of 0 to 10. The ninth question is an open question and answer. The patient is asked to list the three most important causes of the disease. The higher the total score, the greater the threat to the disease.
Self-Efficacy-T1 | T1-baseline
  Cardiac Self-Efficacy Scale have 13 questions in total. The higher the total score, the higher the patient's confidence in dealing with their own heart disease.
Self-Efficacy-T2 | T2-three months later
  Cardiac Self-Efficacy Scale have 13 questions in total. The higher the total score, the higher the patient's confidence in dealing with their own heart disease.
Self-Efficacy-T3 | T3-six months later
  Cardiac Self-Efficacy Scale have 13 questions in total. The higher the total score, the higher the patient's confidence in dealing with their own heart disease.
Anxiety-T1 | T1-baseline
  Beck Anxiety Inventory(BAI) have 21 questions in total. Each question is evaluated with 0-3 points for its severity, with a score of 0- 9 points are normal, 10-18 points are mild anxiety, 19-29 points are moderate anxiety, and 30 points or more are severe anxiety.
Anxiety-T2 | T2-three months later
  Beck Anxiety Inventory(BAI) have 21 questions in total. Each question is evaluated with 0-3 points for its severity, with a score of 0- 9 points are normal, 10-18 points are mild anxiety, 19-29 points are moderate anxiety, and 30 points or more are severe anxiety.
Anxiety-T3 | T3-six months later
  Beck Anxiety Inventory(BAI) have 21 questions in total. Each question is evaluated with 0-3 points for its severity, with a score of 0- 9 points are normal, 10-18 points are mild anxiety, 19-29 points are moderate anxiety, and 30 points or more are severe anxiety.
Cardio-Respiratory Fitness-T1 | T1-baseline
  Six-Minutes Walking Test, 6MWT
Cardio-Respiratory Fitness-T2 | T2-three months later
  Six-Minutes Walking Test, 6MWT
Cardio-Respiratory Fitness-T3 | T3-six months later
  Six-Minutes Walking Test, 6MWT

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsun Chiang, PhD, Principal Investigator — National Defense Medical College, Japan
Locations (1):
- TSGH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No